CLINICAL TRIAL: NCT01614743
Title: A Double-Blinded, Randomized Placebo Controlled Pilot Study Comparing the Efficacy and Safety of IncobotulinumtoxinA Versus Saline Injections to the Cheek Region in Patients With Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DeNova Research (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Principal Investigator, Steven H. Dayan, Medical Director, DeNova Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ROS-INC-12
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IncobotulinumtoxinA (Experimental)
  Interventions: Drug: IncobotulinumtoxinA
- Placebo (Placebo Comparator)
  Interventions: Drug: Bacteriostatic saline

INTERVENTIONS:
Drug: IncobotulinumtoxinA — Experimental injection given at baseline and Week 16
  Arms: IncobotulinumtoxinA
Drug: Bacteriostatic saline — Placebo at baseline, incobotulinumtoxinA at 16 weeks
  Arms: Placebo

SUMMARY:
This is a double-blinded, randomized placebo controlled pilot study comparing the efficacy and safety of incobotulinumtoxinA versus saline injections to the cheek region in patients with rosacea.

The pilot study will enroll and treat a total of 10 subjects who present with rosacea of the cheek area. Upon study entry, subjects will be randomized to receive treatment with incobotulinumtoxinA or bacteriostatic saline to the cheek area. Study treatment will be prepared by an unblinded designee and both Physician Investigator (PI) and subject will remain blinded for the duration of the study. At the 16 week visit, control subjects will enter the rescue arm portion of the study and all study subjects will receive treatment with incobotulinumtoxinA to the cheek areas.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 65 years of age.
2. Subjects presenting with rosacea in the cheek area.
3. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
4. Subjects of childbearing potential must have a negative urine pregnancy test result at Visit 1 and be willing able to use an acceptable method of birth control (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following is documented on the medical history:

   * postmenopausal for at least 12 months prior to study drug administration
   * without a uterus and/or both ovaries
   * has had a bilateral tubal ligation for at least 6 months prior to study drug administration.
   * absence of an other physical condition according to the PI's discretion
5. Willingness and ability to provide written photo consent and adherence to photography procedures (i.e., removal of jewelry and makeup).
6. Willingness and ability to provide written informed consent prior to performance of any study related procedure.

Exclusion Criteria:

1. Subjects who are pregnant, nursing, planning to become pregnant, and/or not using a reliable form of birth control.
2. Subjects with a known allergy or sensitivity to any component of the study medications or anesthesia.
3. Topical or oral rosacea treatments within the past 2 weeks.
4. Subjects with a significant systemic illness or illness localized to the areas of treatment.
5. Botulinum toxin to the face within the past 6 months.
6. Significant concurrent illness such as diabetes, epilepsy, lupus, or congestive heart failure.
7. Concurrent skin condition affecting area to be treated.
8. Prior surgery on the area to be treated within 3 months of initial treatment or during the study.
9. History or evidence of keloids or hypertrophic scarring.
10. Subjects currently using aminoglycoside antibiotics, curare-like agents or other agents that might interfere with neuromuscular function.
11. Subjects with a diagnosis of Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, or any other disease that might interfere with neuromuscular function or current facial palsy.
12. Current history of chronic drug or alcohol abuse.
13. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
14. Subjects who, in the Investigator's opinion, have a history of poor cooperation, non¬compliance with medical treatment or unreliability.
15. Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

REFERENCES:
- See also: DeNova Research Website — http://www.denovaresearch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- IncobotulinumtoxinA at Baseline and Week 16: IncobotulinumtoxinA: Experimental injection given at baseline and Week 16
- Placebo at Baseline, Then incobotulinumtoxinA at 16 Weeks: Bacteriostatic saline: Placebo at baseline, incobotulinumtoxinA at 16 weeks
Period: Overall Study
Arm/Group | IncobotulinumtoxinA at Baseline and Week 16 | Placebo at Baseline, Then incobotulinumtoxinA at 16 Weeks
Started | 4 | 5
Completed | 3 | 5 (Subject in the placebo group (5) also received the treatment (IncobotulinumtoxinA) at Visit 5.)
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 - IncobotulinumtoxinA: Experimental injection given at baseline and Week 16
- Group 2 - Bacteriostatic Saline: Placebo at baseline, incobotulinumtoxinA at 16 weeks
- Total: Total of all reporting groups
Arm/Group | Group 1 - IncobotulinumtoxinA | Group 2 - Bacteriostatic Saline | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 42 [26 to 61] | 53 [47 to 61] | 47 [26 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Rosacea Clinical Score Card
Description: Live rosacea assessment for each side of the face using the Rosacea Clinical Scorecard for clinical assessment.The Rosacea Clinical Scorecard assesses the primary signs and symptoms of rosacea and is graded as absent (0), mild (1), moderate (2) or severe (3).
Time Frame: baseline, 1 week, 4 weeks, 12 weeks, 16 weeks, 17 weeks and 20 weeks
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Group 1 - IncobotulinumtoxinA: IncobotulinumtoxinA: Experimental injection given at baseline and Week 16
- Group 2 - Bacteriostatic Saline: Bacteriostatic saline: Placebo at baseline, incobotulinumtoxinA at 16 weeks
Arm/Group | Group 1 - IncobotulinumtoxinA | Group 2 - Bacteriostatic Saline
Number analyzed (Participants) | 4 | 5
percent change
  % Diff from baseline, Week 1 | -0.63 (0.49) | -0.00063 (0.23)
  % Diff from baseline, Week 4 | -0.65 (0.60) | -0.34 (0.21)
  % Diff from baseline, Week 12 | -0.80 (0.61) | -0.13 (0.13)
  % Diff from baseline, Week 16 | -0.67 (0.48) | -0.51 (0.34)
  % Diff from baseline, Week 17 | -0.83 (0.62) | -0.83 (0.64)
  % Diff from baseline, Week 20 | -1.04 (8.85) | -0.7 (0.53)

2. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Rate of adverse events
Time Frame: baseline, 1 week, 4 weeks, 12 weeks, 16 weeks, 17 weeks and 20 weeks
Measure: Number; unit: participants
Arm/Group | Group 1 - IncobotulinumtoxinA | Group 2 - Bacteriostatic Saline
Number analyzed (Participants) | 4 | 5
participants | 0 | 0

3. Secondary Outcome: Mean Heatherton & Polivy State Self-Esteem (HPSS) Scale Score at Baseline, 1, 4, 12, 16, 17, and 20 Weeks
Description: Self-esteem change will be determined by patient self-evaluation using the Heatherton & Polivy State Self-Esteem (HPSS) Scale.
  Heatherton & Polivy State Self-Esteem (HPSS) Scale includes three facets of self-esteem: Appearance, Performance, and Social The scale has a range of 20-100. A score closer to 100 signifies higher self-esteem, while a score closer to 20 signifies lower seld-esteem.
Time Frame: baseline, 1 week, 4 weeks, 12 weeks, 16 weeks, 17 weeks and 20 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - IncobotulinumtoxinA | Group 2 - Bacteriostatic Saline
Number analyzed (Participants) | 4 | 5
units on a scale
  Baseline | 50.5 (8.19) | 35.2 (10.0)
  Week 1 | 53.0 (11.8) | 36.0 (9.35)
  Week 4 | 53.7 (15.7) | 34.2 (10.1)
  Week 12 | 52.8 (12.6) | 32.2 (7.16)
  Week 16 | 50.3 (11.0) | 34.6 (8.88)
  Week 17 | 52.0 (10.4) | 33.6 (5.32)
  Week 20 | 51.0 (12.2) | 34.2 (8.38)

4. Secondary Outcome: Patient Satisfaction
Description: 4-point categorical assessment of patient satisfaction with treatment.
  1. Highly Satisfied- Optimal cosmetic result
  2. Very Satisfied- Obvious improvement in appearance form the initial condition, but not completely optimal for this subject
  3. Satisfied- Marked improvement in appearance from initial condition
  4. Unsatisfied- The appearance is essentially the same or worse as the original condition.
Time Frame: week 1, 4 weeks, 12 weeks, 16 weeks, 17 weeks and 20 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - IncobotulinumtoxinA | Group 2 - Bacteriostatic Saline
Number analyzed (Participants) | 4 | 5
units on a scale
  Week 1 | 3.0 (0.76) | 3.8 (0.42)
  Week 4 | 2.3 (0.52) | 3.6 (0.52)
  Week 12 | 3.0 (0.0) | 3.3 (0.49)
  Week 16 | 2.7 (0.52) | 3.2 (0.79)
  Week 17 | 2.3 (1.0) | 2.9 (0.32)
  Week 20 | 1.7 (0.52) | 2.2 (0.79)

ADVERSE EVENTS:
Arm/Group | Group 1 - IncobotulinumtoxinA | Group 2 - Bacteriostatic Saline
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
The limitation of this study was a very small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes